CLINICAL TRIAL: NCT05759598
Title: Effect of Respiratory Training Protocols on GH Secretion in the Obese Patient
Brief Title: Effect of Respiratory Training Protocols on GH Secretion in Obesity (ALRESPGHOB)
Acronym: ALRESPGHOB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of hormonal responses (GH) in response to the respiratory training protocols in the three subjects tested.
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01C020
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Obesity
Keywords: Growth hormone; Insulin-like growth factor; Training of respiratory muscles
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CTRL) (Other)
  Interventions: Other: Rehabilitation protocol + guided spontaneous breathing exercises
- Experimental group (RMT) (Experimental)
  Interventions: Other: Rehabilitation protocol + specific respiratory muscle training program

INTERVENTIONS:
Other: Rehabilitation protocol + guided spontaneous breathing exercises — Standard integrated metabolic rehabilitation protocol + guided spontaneous breathing exercises
  Arms: Control group (CTRL)
Other: Rehabilitation protocol + specific respiratory muscle training program — Standard integrated metabolic rehabilitation protocol + specific respiratory muscle training program according to the protocol recently proposed by Spengler et al. (Wuthrich et al., 2015; Schaer et al., 2018), adapted according to the baseline characteristics of the respiratory function of the subjects
  Arms: Experimental group (RMT)

SUMMARY:
The study's primary objective is to evaluate the acute and chronic (3 weeks) effects of two respiratory training protocols in obese adolescents (performed during a period of hospitalization for a body weight reduction program), with different characteristics and mechanisms of action, on GH and IGF-I secretion. The definition of the protocols is based on what has been observed by recent studies conducted on healthy people (Wuthrich et al., 2015; Schaer et al., 2018) and on patient populations in which respiratory dysfunction is a primary or secondary component of the pathology (Calcaterra et al., 2014; Pomidori et al., 2009). All planned interventions are safe and are adapted to the obese patient.

Project objectives are:

* assessment of GH-IGF-I responses (baseline), during the first training session of the respiratory muscles conducted in the first days of hospitalization of the patients in the clinic
* assessment of GH-IGF-I responses (post), during the last training session of the respiratory muscles conducted at the end of the three weeks of each training session

DETAILED DESCRIPTION:
Materials and methods:

Subjects The study provides for the recruitment of 20 obese boys/young adults aged between 14 and 30 years old hospitalized at the Division of Auxology and the Division of Metabolic Diseases, Istituto Auxologico Italiano, S. Giuseppe Hospital, Piancavallo (VB).

Criteria for inclusion in the study group are:

1. BMI standard deviation score (SDS)>2 for patients < 18 years and BMI>35 for patients aged>18 years;
2. absence of structured physical activity programs (regular activity for more than 120 minutes/week) during the 6 months preceding the study;
3. absence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal, or musculoskeletal pathologies contraindicated for carrying out the tests.

Materials and methods:

During the first respiratory training session (basal) and at the end of the three weeks of hospitalization (post) for an integrated metabolic rehabilitation program at the Division of Auxology (patients aged < 18 years) and Division and Metabolic Diseases (adults) a blood sample is taken from each subject to determine the circulating levels of GH (total and isoforms 20 kDa and 22kDa) and cortisol in pre-training conditions and at times 0 ' (immediately at the end), +15', +30' and +60' (IGF-I levels are determined only in pre-workout conditions and immediately at the end). Blood samples taken after training are carried out by needle cannula during a saline infusion, to reduce the number of venipunctures. Lactate levels are determined by earlobe puncture in basal conditions, immediately at the end of the training session, and repeated every 2 minutes, until the peak value is reached.

In baseline conditions and at the end of the 3 weeks of respiratory training, body composition is evaluated (by impedance analysis), the maximum force developed during voluntary isometric contraction of the extensor and flexor muscles of the lower limb (by dynamometer), and spirometry is performed for the assessment of maximal lung capacity.

Respiratory muscle training protocol:

The recruited subjects are randomly divided into two homogeneous groups in terms of the number and basic characteristics of the subjects. A control group (CTRL) carries out the standard integrated metabolic rehabilitation protocol with the addition of guided spontaneous breathing exercises lasting about 20 minutes per session for 12 sessions.

An experimental group (RMT) carries out, in addition to the standard integrated metabolic rehabilitation protocol, a specific respiratory muscle training program according to the protocol recently proposed by Spengler et al. (Wuthrich et al., 2015; Schaer et al., 2018), adapted according to the baseline characteristics of the respiratory function of the subjects. The protocol includes 12 interval breathing training sessions, divided into 3 weeks (4 sessions/week) each lasting a total of about 12 minutes. Each respiratory training session includes 6 1-minute "sprint" breathing intervals followed by 1 minute of recovery. During the sprint intervals, the subjects breathe through a dedicated SpiroTiger instrument (Idiag AG, Fehraltorf, Switzerland) with the addition of a resistance (Schaer et al., 2018) which allows normocapnic hyperpnea against resistance. Subjects are asked to breathe at a respiratory rate of 25-30 breaths/minute with a constant tidal volume corresponding to approximately 60% of forced vital capacity. The target frequency is adjusted on an individual basis and is defined during the initial familiarization trials.

ELIGIBILITY:
Inclusion Criteria:

* BMI standard deviation score (SDS) > 2 for subjects aged < 18 years and BMI > 35 for patients aged >18 years;
* absence of structured physical activity programs (regular activity for more than 120 minutes/week) during the 6 months preceding the study;
* absence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal, or musculoskeletal pathologies contraindicated for carrying out the tests.

Exclusion Criteria:

* age < 14 years and > 30 years;
* presence of structured physical activity programs (regular activity for more than 120 minutes/week) during the 6 months preceding the study;
* presence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal, or musculoskeletal pathologies contraindicated for carrying out the tests.

Ages: 14 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Growth hormone (GH) | Baseline, 0, 15, 30 and 45 minutes after Intervention and 3 weeks after intervention
  Change in plasma concentration of growth hormone
Insulin-like growth factor (IGF-I) | Baseline and 0 minutes after Intervention
  Change in plasma concentration of insulin-like growth factor

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Site Piancavallo, Oggebbio, Verbania, Italy